CLINICAL TRIAL: NCT05466799
Title: An Open-label, Multi-centre, Randomized Study of TaRgeted Intratumoural Placement of P-32 (OncoSil™) in Addition to FOLFIRINOX Chemotherapy vs FOLFIRINOX Alone in Patients With Unresectable Locally Advanced Pancreatic Adenocarcinoma.
Brief Title: FOLFIRINOX Versus OncoSil™ in Addition to FOLFIRINOX in Patients With Locally Advanced Pancreatic Adenocarcinoma
Acronym: TRIPP-FFX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OncoSil Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCO01P04
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Leucovorin; Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFIRINOX Chemotherapy (Active Comparator): Subjects in Arm A will receive up to 12 cycles of Standard Of Care FOLFIRINOX chemotherapy
  Interventions: Drug: FOLFIRINOX chemotherapy
- OncoSil™ in addition to FOLFIRINOX Chemotherapy (Experimental): Subjects in Arm B will be implanted with the OncoSil™ device in addition to up to 12 cycles of Standard Of Care FOLFIRINOX chemotherapy
  Interventions: Drug: FOLFIRINOX chemotherapy; Device: OncoSil™

INTERVENTIONS:
Drug: FOLFIRINOX chemotherapy — Standard Of Care Chemotherapy regimen for treatment of Locally Advanced Pancreatic cancer
  Other Names: Folinic Acid, 5-FU, Oxaliplatin, Irinotecan
Device: OncoSil™ — Implantation of OncoSil 32P microparticles into the Pancreatic Tumour under EUS guidance
  Other Names: Phosphorous-32 microparticles
  Arms: OncoSil™ in addition to FOLFIRINOX Chemotherapy

SUMMARY:
The purpose of the study is to assess the safety and efficacy of OncoSil™ when given in addition to standard FOLFIRINOX chemotherapy for treatment of Locally Advanced Pancreatic Cancer

DETAILED DESCRIPTION:
Patients with Locally Advanced Pancreatic Cancer who have not received prior treatment to their pancreatic cancer will be informed about the study and the potential risks and benefits. After providing informed consent patients will undergo a 3 week screening period to confirm eligibility for the study. Patients who meet all eligibility criteria will be randomised 1:1 to either the control arm of up to 12 cycles of standard of care FOLFIRINOX chemotherapy or implantation of OncoSil™ in addition to the same FOLFIRINOX chemotherapy regimen. Patients will be followed for side side effects and palliative benefits during 4-8 weekly study visits and the objective efficacy of the treatment will be assessed by CT scans every 8 weeks. Quality of Life will be measured on various time-points using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven adenocarcinoma of the pancreas.
2. Unresectable locally advanced pancreatic adenocarcinoma according to NCCN 2021 guidelines.Staging and unresectability must be confirmed by central review of the baseline CT scan.
3. Pancreatic target tumour diameter of < 7.0 cm (longest axis), as qualified by the central reading centre.
4. Karnofsky Performance Status ≥ 70
5. ≥ 18 years of age at screening.
6. Considered fit to commence first-line standard FOLFIRINOX chemotherapy:

   i) Adequate renal function: serum creatinine less than 1.5 x upper limit of normal (ULN).

   ii) Adequate liver function: serum liver transaminases ≤ 3 x ULN and serum bilirubin ≤ 1.5 x ULN*.

   *For study participants with recent biliary obstruction treated by drainage (e.g. stent), serum bilirubin of > 1.5 x ULN will be accepted for study entry provided that serial levels demonstrate clear improvement. In addition, chemotherapy should not be commenced until serum bilirubin is ≤ 1.5 x ULN.

   iii) Adequate bone marrow function: white blood cells (WBCs) ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, haemoglobin ≥ 9 g/dL, and platelets ≥ 100,000/mm3 iv) UGT1A1 polymorphism and DPD deficiency test performed and dose reductions applied as per local institutional practice.
7. Provide signed Informed Consent.
8. Willing and able to complete study procedures within the study timelines.
9. Life expectancy of at least 3 months at the time of screening as judged by the investigator.
10. Treated with or eligible to commence prophylactic treatment with a proton-pump inhibitor prior to implantation, and to continue to receive treatment for at least 6 months post implantation.
11. Not pregnant, and if of childbearing potential, agrees to use adequate birth control (hormonal or barrier method of birth control or abstinence) prior to study entry and during the study and agrees not to donate sperm or ova, for the duration of the study and 12 months post implantation of the investigational device.

Exclusion Criteria:

1. Evidence of distant metastases, based on review of baseline CT scan.
2. More than one pancreatic tumour lesion.
3. Any prior radiotherapy or chemotherapy for pancreatic cancer.
4. Pregnant or lactating.
5. In the opinion of the investigator, EUS-directed implantation posing undue study subject risk. This includes:

   i) where previous EUS-FNA was considered technically too difficult to perform; ii) imaging demonstrates multiple collateral vessels surrounding or adjacent to the target tumour within the pancreas; iii) presence (or significant risk) of varices near to the target tumour. Note: The feasibility of implantation of the target tumour and assessment of risk can be repeated at any time between Screening Visit 1 and the implantation date. If any of the above risk features becomes apparent following subject screening and/or enrolment prior to and including at the time of OncoSil™ treatment, the patient should remain in the study but the implantation should be deferred or cancelled.
6. History of malignancy, treated or untreated, within the past five years whether or not there is evidence of local recurrence or metastases, with the exception of basal cell carcinoma of the skin and cervical carcinoma in situ.
7. Evidence of radiographic invasion into stomach or duodenum (if not certain, confirmation must be obtained prior to enrolment).
8. A known history of hypersensitivity to silicon or phosphorous, or any of the OncoSil™ components.
9. Any other health condition that would preclude participation in the study in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Through study completion, an average of 18 months
  The primary analysis for safety of OncoSil™ is defined by the Adverse Event profile
Local Disease Control Rate (LDCR) at 16 Weeks | 16 weeks after initiation of FOLFOX chemotherapy
  The LDCR at Week 16 will be summarised as a count and proportion of subjects with Local Disease Control at 16 Weeks

SECONDARY OUTCOMES:
Local Progression Free Survival (LPFS), within the pancreas | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  Local Progression Free Survival (LPFS) is defined as the time from enrolment to the date of the radiological scan used to determine local tumour progression or date of death from any cause, whichever comes first.
Progression Free Survival | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  Progression free survival (PFS) is defined as the time from enrolment to the date of tumour progression or of recurrence (in case of complete response (CR) or resection of the primary pancreatic tumour), or death from any cause, whichever comes first.
Time to symptomatic progression | From date of enrolment until the date of symptomatic progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  Time to symptomatic progression is defined as the time between enrolment and worsening of cancer related symptoms as measured by the symptoms domains of QLQ-C30/PAN26
Clinical Benefit Response | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  Clinical Benefit Response is a composite endpoint consisting of weight, Performance Status and pain score and will be derived at 4 weekly intervals.The frequency and percentage of subjects with a clinical benefit response will be summarised
CA 19-9 response | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  CA 19-19 response will be defined as ≥ 50% decline from baseline and ≥ 90% decline from baseline and return to normal range respectively. Subgroups will be created for study subjects with CA 19-9 > ULN at baseline.
Overall Survival | Through study completion, an average of 18 months
  Overall survival (OS) is the time from enrolment to the date of death from any cause.
Patient Reported Outcomes | Through study completion, an average of 18 months
  EQ-5D, EORTC QLQ-C30 and PAN26 will be analyses per their validated methodology
Pain Scores | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  NRS and QLC-PAN26
Weight loss | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  weight will be assessed at all applicable study visits
Tumour response | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  RECIST 1.1 per central review
Surgical resection rate | Through study completion, an average of 18 months
  assessment of rate of secondary R0/R1 resection
Target Tumour Volumetric Change | From date of enrolment until the date of first documented local progression or date of death from any cause, whichever came first, assessed up to 7 months after last enrolled patient
  A central reading centre will analyse all CT scans to measure target tumour volume changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Milella, MD, PhD, Principal Investigator — University Hospital of Verona; Giuseppe Malleo, MD, PhD, Principal Investigator — University Hospital of Verona
Locations (17):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Epworth Healthcare, Richmond, Victoria
- AZ Maria Middelares, Ghent, Belgium
- Italy (2):
  - San Camillo Forlanini, Rome
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octobre, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (5):
  - Guy's Hospital, London
  - Imperial College, London
  - The Christie Hospital/Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared on an individual basis to study investigators subject to review and approval from the study publication steering committee
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After the release of the primary study publication
Access Criteria: Request should be made to the chair of the publication steering committee with specification of the proposed analysis and the required IPD